CLINICAL TRIAL: NCT05691569
Title: Efficacy of Doll Therapy in the Control of Behavioral and psychologIcal Symptoms of Dementia in Acute Geriatric Inpatients: the AGITATE Study.
Brief Title: Efficacy of Doll Therapy in the Dementia in Acute Geriatric Inpatients
Acronym: AGITATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Patrizia D'Amelio, Full professor, head of the geriatric and Geriatric rehabilitation Service, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: agitate
Record Dates: First submitted 2022-11-29; First posted 2023-01-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled open label trial with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- doll therapy (Experimental): The doll used in the study is the "empathy doll"; these dolls are designed to obtain an optimal interaction with patients and to arouse empathy
  Interventions: Other: doll therapy
- non anthropomorphic object (Other): non- anthropomorphic soft object
  Interventions: Other: doll therapy

INTERVENTIONS:
Other: doll therapy — empathy dolls

SUMMARY:
Summary. Behavioral and psychological symptoms of dementia (BPSD) represents a huge emotional stress and an important burden for the patients and the caregivers severely reducing their quality of life. BPSD worsen during hospitalization and require the administration of psychotropic drugs that are often insufficient to control the symptoms, and may cause severe adverse events.

The investigators propose the use of empathy dolls in order to reduce BPSD and in particular agitation and aggressiveness in acute geriatric in-patients affected by moderate to severe forms of dementia.

The use of doll therapy in the clinical routine will allow to reduce the use of psychotropic drugs, shorten hospitalization, reduce professional and family caregiver burden improving patients' and families' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age ≥65 years
* diagnosis of dementia moderate to severe Clinical Dementia Rating scale (CDR) ≥2
* presence of agitation and/or aggressiveness
* manual and visual abilities sufficient in order to interact with the doll.

Exclusion Criteria:

* age <65 years;
* refuse to participate;
* mild forms of dementia (CDR<2);
* contraindication for DT as experience of mournful or traumatic events related to parental experience;
* life expectancy lower than 3 months;
* infectious diseases requiring isolation;
* negative interaction with the doll,
* presence of delirium.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
agitation and aggressiveness within hospital | baseline and hospital discharge discharge (up to one week)
  measured by Pittsburgh Agitation Scale (PAS). the score ranges between 0 to 16 on the PAS the higher score means the higher agitation
behavioural and psychological symptoms of dementia | baseline, discharge (up to one week)
  Neuro Psychiatic Inventory (NPI). The NPI total score ranges from 0 to 144, higher scores means more severe and frequent behavioural and psycological symptoms of dementia
agitation and aggressiveness outside hospital | baseline, 1 and 4 weeks after discharge
  Cohen Mansfield Inventory scale (CMAI). the score ranges betwen 0 and 203, with higher scores indicating more agitation

SECONDARY OUTCOMES:
incidence of delirium | every day during hospital stay (up to one week)
  measured by the Confusion Assessment Method (CAM) scale. For a diagnosis of delirium by CAM, the patient must display:
  1. Presence of acute onset and fluctuating discourse AND
  2. Inattention AND EITHER
  3. Disorganized thinking OR
  4. Altered level of consciousness
patients' quality of life | baseline and 4 weeks after discharge
  by the use of the AD-5D Dementia Utility Instrument, the scales scores between -1 to 1, the highest score indicate the better quality of life
family caregivers' quality of life | baseline and 4 weeks after discharge
  by the EuroQoL 5-Dimensions 5 level versions. the scale scores from 5 to 25 the highest the score the lowest the quality of life
professional caregiver burden | baseline and at hospital discharge (up to one week)
  Staff Stress Measure Dementia Care (SSMDC). The scale comprised the following 27 items producing a five-factor solution: Frustrated empathy; difficulties understanding and interpreting; balancing competing needs; balancing emotional involvement; and lack of recognition.
family caregiver burden | baseline and 4 weeks after discharge
  Caregiver Burden Inventory (CBI) scale. The Caregiver Burden Inventory comprises 24 closed questions divided into five dimensions: time-dependence, developmental, physical, social and emotional burden. There are five items in each dimension except for physical burden, which has four items dedicated to. Each item is given a score between 0 (not at all descriptive) and 4 (very descriptive), where higher scores indicate greater caregiver burden; there are no cut-off points for classifying burden. Therefore, total scores for factors one, two, four and five can range from zero to 20. An equivalent score for physical burden can be obtained by multiplying the sum of items in this dimension by 1.25

CONTACTS AND LOCATIONS:
Locations (1):
- geriatric and Geriatric Rehabilitation Unit, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin-Garcia A, Corregidor-Sanchez AI, Fernandez-Moreno V, Alcantara-Porcuna V, Criado-Alvarez JJ. Effect of Doll Therapy in Behavioral and Psychological Symptoms of Dementia: A Systematic Review. Healthcare (Basel). 2022 Feb 23;10(3):421. doi: 10.3390/healthcare10030421. PMID 35326899
- [Background] Molteni V, Vaccaro R, Ballabio R, Ceppi L, Cantu M, Ardito RB, Adenzato M, Poletti B, Guaita A, Pezzati R. Doll Therapy Intervention Reduces Challenging Behaviours of Women with Dementia Living in Nursing Homes: Results from a Randomized Single-Blind Controlled Trial. J Clin Med. 2022 Oct 24;11(21):6262. doi: 10.3390/jcm11216262. PMID 36362489
- [Background] James IA, Reichelt K, Shirley L, Moniz-Cook E. Management of Agitation in Behaviours That Challenge in Dementia Care: Multidisciplinary Perspectives on Non-Pharmacological Strategies. Clin Interv Aging. 2023 Feb 18;18:219-230. doi: 10.2147/CIA.S399697. eCollection 2023. PMID 36843632
- [Background] Peng Y, Liu Y, Guo Z, Zhang Y, Sha L, Wang X, He Y. Doll therapy for improving behavior, psychology and cognition among older nursing home residents with dementia: A systematic review and meta-analysis. Geriatr Nurs. 2024 Jan-Feb;55:119-129. doi: 10.1016/j.gerinurse.2023.10.025. Epub 2023 Nov 19. PMID 37980780
- [Background] Santagata F, Massaia M, D'Amelio P. The doll therapy as a first line treatment for behavioral and psychologic symptoms of dementia in nursing homes residents: a randomized, controlled study. BMC Geriatr. 2021 Oct 12;21(1):545. doi: 10.1186/s12877-021-02496-0. PMID 34641791